CLINICAL TRIAL: NCT05753241
Title: Hospital of Chengdu University of Traditional Chinese Medicine
Brief Title: the Relationship Between Allergic Rhinitis and the Risk of Symptom in Patients With Mild COVID-19
Status: Completed | Type: Observational
Sponsor: qinxiu zhang (Other)
Responsible Party: Sponsor-Investigator, qinxiu zhang, Professor, School of Clinical Medicine, Chengdu University of Traditional Chinese Medicine, Chengdu University of Traditional Chinese Medicine
Organization: Chengdu University of Traditional Chinese Medicine (Other)
Other Study IDs: CDUTCM20230301
Record Dates: First submitted 2023-03-01; First posted 2023-03-03 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: COVID-19; Allergic Rhinitis
Keywords: allergic rhinit; sublingual immunotherapy; the symptoms after COVID-19 infection; Odds ratio
MeSH Terms: conditions — COVID-19; Rhinitis, Allergic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- healthy group (HG): Participants were grouped according to their basic conditions without any intervention
  Interventions: Other: no intervention
- allergen immunotherapy group (AIT): Participants were grouped according to their basic conditions without any intervention
  Interventions: Other: no intervention
- allergic rhinitis group (ARG): Participants were grouped according to their basic conditions without any intervention
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — It's only observational study. No interventions.

SUMMARY:
At present, most studies mainly focussed on severe patients, and there was no comparison of symptom differences between AR patients and healthy people with mild infection to evaluate the symptoms of AR patients during infection and to provide preventive treatment in advance. So this experiment was designed.

DETAILED DESCRIPTION:
After the end of this large-scale infection, the investigators analyzed the re-diagnosis of patients with allergic rhinitis (AR) at the Otolaryngology Clinic, and found significant differences in symptoms between AR and non-AR patients. AR patients had more serious nasal and pharyngeal symptoms. In previous studies on the correlation between allergic diseases and COVID-19 infection, AR was found to be a protective factor to reduce COVID-19 infection and the risk of severe disease . In contrast, a cohort study in South Korea found that AR worsened COVID-19 infection . These studies mainly focussed on severe patients, and there was no comparison of symptom differences between AR patients and healthy people with mild infection.

Allergy may lead to the overall damage of nasal mucosa due to the mechanical and immune defense function of the virus. Immunotherapy will significantly reduce the number and severity of upper respiratory tract infections (including children's common cold). The investigators hypothesized that AR is more likely to aggravate symptoms after infection, while allergen immunotherapy （AIT） may reduce the risk of symptoms as a protective factor for symptoms after AR virus infection. Therefore, the investigators conducted a retrospective analysis on the risk of symptoms after COVID-19 infection in patients with AR, and compared the difference of symptoms after COVID-19 infection in patients with AIT and non-AIT AR.

ELIGIBILITY:
Inclusion Criteria:

* all participants completed at least one antigen or nucleic acid test and the results were positive.
* the diagnoses of AR met the international diagnostic standards for AR. The participants had obvious clinical symptoms and the allergen test was positive.

Exclusion Criteria:

* suspected new infected person with symptoms（ no antigen or nucleic acid test and the results were nagetive ）
* Participants requiring ICU admission after COVID-19 infection-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study period will include all patients attending the ENT outpatient clinic (AR and NO-AR) from December 1, 2022 to December 1, 2023
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Actual)
Dates: Start 2022-11-10 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-06-22 (Actual)

PRIMARY OUTCOMES:
post-infection symptoms（pharyngeal symptoms；Systemic symptoms； Gastrointestinal symptoms；Olfactory and gustatory dysfunction；Severe symptoms） | The first day after COVID-19 infection
  pharyngeal symptoms: dry throat, itchy throat, sore throat, cough, expectoration; Systemic symptoms: fever, headache, fatigue, cold limbs; Gastrointestinal symptoms: diarrhea, constipation; Olfactory and gustatory dysfunction: hypoosmia, hypogustia; Severe symptoms: chest tightness, pant, palpitation, convulsion, coma.
hospitalization rate | The first day after COVID-19 infection
  The probability of needing hospital treatment after infection

CONTACTS AND LOCATIONS:
Overall Officials: qinxiu zhang, Dr., Principal Investigator — Chengdu University of Traditional Chinese Medicine
Locations (1):
- Hospital of Chengdu University of Traditional Chinese Medicine, Chengdu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zhang S, Liu C, Liu Q, He X, Fu Q, Chen X, Jin X, Chen Z, Yang X, Zhang Q, Li X. The relationship between sublingual immunotherapy for allergic rhinitis and the risk of symptoms in patients with COVID-19 infection. Hum Vaccin Immunother. 2023 Aug 1;19(2):2236538. doi: 10.1080/21645515.2023.2236538. PMID 37530139
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC10399475/